CLINICAL TRIAL: NCT03899298
Title: Safety and Clinical Outcomes Study: Amniotic and Umbilical Cord Tissue Administration for Orthopedic, Neurologic, Urologic, Autoimmune, Renal, Cardiac and Pulmonary Conditions
Brief Title: Safety and Clinical Outcomes With Amniotic and Umbilical Cord Tissue Therapy for Numerous Medical Conditions
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: R3 Stem Cell (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #2018/10/11
Record Dates: First submitted 2019-03-27; First posted 2019-04-02 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-03

CONDITIONS: Orthopedic Disorder; Neurologic Disorder; Urologic Diseases; Erectile Dysfunction; Autoimmune Diseases; Renal Failure; Renal Insufficiency; Kidney Diseases; Cardiac Event; Cardiomyopathies; CHF; Pulmonary Disease; COPD; Alzheimer Disease; Stroke; Neuropathy;Peripheral; Arthritis
Keywords: stem cell therapy; umbilical stem cells; amniotic stem cells; stem cells; regenerative medicine; r3 stem cell; perinatal tissue; placenta stem cell
MeSH Terms: conditions — Musculoskeletal Diseases; Nervous System Diseases; Urologic Diseases; Erectile Dysfunction; Autoimmune Diseases; Renal Insufficiency; Kidney Diseases; Cardiovascular Diseases; Cardiomyopathies; Lung Diseases; Pulmonary Disease, Chronic Obstructive; Alzheimer Disease; Stroke; Neuritis; Arthritis

STUDY DESIGN:
Intervention Model Description: The study will be ongoing for patient inclusion and data acquisition. Patients will be separated into one of seven categories including: Orthopedic, Neurologic, Urologic, Autoimmune, Renal, Cardiac and Pulmonary Conditions. The treatments will not be randomized or blinded. This is a partially patient funded study. The study has been approved by an Alion accredited Institutional Review Board, Solutions IRB as of March 2019.
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Amniotic and Umbilical Cord Tissue for Autoimmune Conditions (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for autoimmune conditions. Outcomes will be compared to the literature results of the current gold standard for several conditions.
  Interventions: Biological: Amniotic and Umbilical Cord Tissue Procedure
- Amniotic and Umbilical Cord Tissue for Orthopedic Conditions (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for orthopedic conditions. Outcomes will be compared to the literature results of the current gold standard for several conditions.
  Interventions: Biological: Amniotic and Umbilical Cord Tissue Procedure
- Amniotic and Umbilical Cord Tissue for Neurologic Conditions (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for neurologic conditions. Outcomes will be compared to the literature results of the current gold standard for several conditions.
  Interventions: Biological: Amniotic and Umbilical Cord Tissue Procedure
- Amniotic and Umbilical Cord Tissue for Urologic Conditions (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for urologic conditions. Outcomes will be compared to the literature results of the current gold standard for several conditions.
  Interventions: Biological: Amniotic and Umbilical Cord Tissue Procedure
- Amniotic and Umbilical Cord Tissue for Cardiac Conditions (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for cardiac conditions. Outcomes will be compared to the literature results of the current gold standard for several conditions.
  Interventions: Biological: Amniotic and Umbilical Cord Tissue Procedure
- Amniotic and Umbilical Cord Tissue for Renal Conditions (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for renal conditions. Outcomes will be compared to the literature results of the current gold standard for several conditions.
  Interventions: Biological: Amniotic and Umbilical Cord Tissue Procedure
- Amniotic and Umbilical Cord Tissue for Pulmonary Conditions (Experimental): Purpose is to evaluate an amniotic and umbilical cord stem cell rich tissue substance for pulmonary conditions. Outcomes will be compared to the literature results of the current gold standard for several conditions.
  Interventions: Biological: Amniotic and Umbilical Cord Tissue Procedure

INTERVENTIONS:
Biological: Amniotic and Umbilical Cord Tissue Procedure — Amniotic and Umbilical Cord Cell Therapy with protocols dependent on the patient condition. Protocols include options for IV, Injection, Intranasal and/or Nebulizer.
  Other Names: Amniotic and Umbilical Cord Tissue Infusion; Amniotic and Umbilical Cord Tissue Nebulizer; Amniotic and Umbilical Cord Tissue Injection; Amniotic and Umbilical Cord Tissue Intranasal

SUMMARY:
To determine the safety and efficacy of Amniotic and Umbilical Cord Tissue for the treatment of the following condition categories: Orthopedic, Neurologic, Urologic, Autoimmune, Renal, Cardiac and Pulmonary Conditions. The hypotheses are that the treatments are not only extremely safe, but also statistically beneficial for all conditions. Outcomes will be determined by numerous valid outcome instruments that compile general quality of life information along with condition-specific information as well.

DETAILED DESCRIPTION:
The study will be ongoing for patient inclusion and data acquisition. Patients who have Orthopedic, Neurologic, Urologic, Autoimmune, Renal, Cardiac and Pulmonary Conditions will be included.

The study has been approved by an Alion accredited Institutional Review Board, Solutions IRB, as of March 2019.

Depending on the condition, patients may receive a series of therapies via one or more of the following methods: intravenous, injection, intra-nasal and/or nebulizer. R3 has several "best practice" therapy protocols that participating practices will follow. Should a patient have conditions that fall into more than one condition category, he or she can still be included with the protocols being received for each condition(s).

Here is a specific administration for each condition category:

1. Orthopedic Condition = Injection
2. Neurologic Disease = IV Infusion and Intranasal Procedure. The exception is with Peripheral Neuropathy, where participants receive a series of injections along with an IV Infusion Procedure.
3. Urologic = Injection
4. Autoimmune = IV Infusion
5. Cardiac = IV Infusion
6. Pulmonary = IV Infusion plus Nebulizer
7. Renal = IV Infusion

Pre, Intra and Post procedure data acquisition will occur at various time frames up to 10 years. Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months, 36 months and then on average each year, up to 10 years. Patients will pay for procedures, and no randomization will occur.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and over.
2. Ability to attend follow up visits or at least converse on phone or complete email follow up forms.
3. Competent to understand the study protocol and provide voluntary informed consent.
4. Patients with any of the following conditions: Arthritis (Degenerative, Rheumatoid, Psoriatic, Lupus, Gout), Sports or Overuse Injuries (e.g. Rotator Cuff injury, Tennis Elbow), Chronic Kidney Disease (may be on dialysis), Back/Neck Pain, Erectile Dysfunction, Peyronie's Disease, Alzheimer's Disease, Parkinson's Disease, Neuropathy, Post-Stroke, Post-Concussion Syndrome, COPD, Emphysema, Pulmonary Fibrosis, Post myocardial infarction (at least 6 months out), Cardiomyopathy, Congestive Heart Failure.

Exclusion Criteria:

1. Active Cancer
2. Pregnancy, Lactating
3. Severe Clotting disorder
4. Myocardial Infarction less than six months ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2024-03-20 (Estimated); Study Completion 2029-03-20 (Estimated)

PRIMARY OUTCOMES:
Disabilities of Arm, Shoulder, Hand Questionnaire (DASH) | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  Upper Extremity Outcome Instrument
Sexual Health Inventory for Men Questionnaire (SHIM) | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  Erectile Function Questionnaire. Scoring exists from 0 to 25. The lower the score, the more severe the Erectile Dysfunction.
Kidney Disease and Quality of Life Questionnaire (KDQOL) | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  Renal Function Outcome Instrument. Raw, precoded numeric values for 36 items are transformed linearly to a 0 to 100 range, with higher scores reflecting better quality of life.
Assessment of Quality of Life Questionnaire (AQOL) | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  General Health Outcome Instrument. Each instrument is used to derive a simple psychometric score for health related quality of life (HRQoL) and to provide profile scores on the different dimensions or items of the descriptive systems. The score is derived by adding the unweighted response order of each question, with a lower score denoting a better quality of life.
Clinical Chronic Obstructive Pulmonary Disease Questionnaire | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  COPD Outcome Instrument. Items are scored on a Likert scale (range 0-60). Higher scores indicate a worse health status.
Mini Mental State Examination (MMSE) | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  Memory Outcome Instrument. The maximum MMSE score is 30 points. The lower the score, the more severe the dementia.
O'Leary/Sant Questionnaire | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  Voiding and Pain Indices. Possible score of 0-20 with higher scores denoting better function.
Oswestry Low Back Pain Disability Questionnaire | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  Low Back Pain Outcome Instrument. Possible score of 0-100 with lower scores denoting better function.
Western Ontario and McMaster Osteoarthritis Index (WOMAC) | Follow up time-frames will measure changes occurring from baseline post procedure at 1 month, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 36 months, 48 months, 60 months, 72 months, 84 months, 96 months, 108 months and 120 months.
  Arthritis Outcome Instrument. Individual question scores are then summed to form a raw score ranging from 0 (worst) to 96 (best).

CONTACTS AND LOCATIONS:
Overall Officials: David Greene, MD, MBA, Study Director — R3 Stem Cell

IPD SHARING:
Plan to Share IPD: No
Data will be blinded and password protected. Research publications will be produced for medical journals. Participating Investigators will have password protected access only.

REFERENCES:
- See also: R3 Stem Cell — http://r3stemcell.com